CLINICAL TRIAL: NCT04929821
Title: UNITY-B A Prospective, Multicentric, Single-arm Study to Evaluate the Safety and Efficacy of the UNITY-B Biodegradable Balloon-Expandable Biliary Stent System in Subjects With Biliary Strictures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: QualiMed Innovative Medizinprodukte GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUA-CLI-UN-01/QM-IS-UTB-035
Record Dates: First submitted 2020-08-20; First posted 2021-06-18 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Biliary Obstruction; Bile Duct Stricture; Bile Duct Diseases
MeSH Terms: conditions — Bile Duct Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Device Treated Group (Other): Treated with the study device, UNITY-B Biodegradable Balloon-Expandable Biliary Stent System.
  Interventions: Device: Biliary Duct Stenting

INTERVENTIONS:
Device: Biliary Duct Stenting — UNITY-B Balloon-expandable Biodegradable Biliary Stent deployment in obstructed biliary ducts.

SUMMARY:
STUDY TYPE: Feasibility study STUDY DESIGN: Prospective, multicenter, single-arm, open-label PRIMARY OBJECTIVE The primary objective is to assess safety of the UNITY Balloon-expandable Biodegradable Biliary Stent System SECONDARY OBJECTIVES Clinical /Technical /Procedural success, Quality of Life improvement, biodegradation rate

DETAILED DESCRIPTION:
RATIONALE (STUDY PURPOSE) Recent publications report the experience with temporary placement of self-expanding metallic stents (SEMS) in benign biliary strictures, which could offer several advantages over conventional plastic biliary stents. Removability can be complicated when there is tissue ingrowth through uncovered portions of the biliary SEMS.

Use of a biodegradable stent would eliminate procedural risk and expense associated with stent removal. In addition, a stent made of highly biocompatible material may be less prone to induce hyperproliferative damage to the ductal system than would plastic or metal stents. For biliary applications, biodegradable stents have been evaluated in several in-vitro and animal studies that proved the stents for being safe and well tolerated. They provided an adequate radial force and resulted in complete stricture resolution within several months. The stents did not show any signs of biliary hyperplasia or integration in the epithelium. Moreover, they seem to have a self-clearing effect on attached biofilm as the outer layer sloughs during the degradation process similarly to the exfoliation of human skin. Also, the stent could be removed from the bile duct, thus offering the possibility of extraction if necessary, at various times after implant.

Therefore, the aim of this clinical study is to evaluate the safety and the efficacy of the UNITY-B Biodegradable Balloon Expandable Biliary Stent System for draining obstructed biliary ducts to improve bile flow in patients suffering under biliary strictures accompanied by jaundice and pruritus or to maintain good clinical status for patients already drained by PTBD or primary stenting.

STUDY DEVICE The UNITY Balloon-expandable Biodegradable Biliary Stent System is comprised of two main components: a balloon-expandable, biodegradable hybrid stent and an over-the-wire balloon catheter delivery system. The UNITY-B System provides a means of safely advancing the stent to the desired location within the common bile duct and, once in position, the stent is deployed by inflating the balloon. The balloon expands to the nominal diameter under nominal pressure. The process in which the UNITY- B stent degrades is through hydrolysis. Implantation is endoscopally guided (ERCP) and stent advancement and deployment by virtue of a guide wire and balloon catheter. In cases of altered anatomy this device can be used for percutaneous transhepatic access as well.

POPULATION Patients with biliary strictures and suffer under jaundice associated with tea color urine, pale stool and pruritus. Biliary drainage relieves both and improves related symptoms like anorexia, diarrhea, and disturbed sleep pattern and leads to improved quality of life. Patient with previous PTBD or stenting who need secondary stenting for prolonged good clinical status.

PRIMARY ENDPOINT (Safety) The primary safety endoint is the proportion of subjects experiencing biliary and procedural complications (post-ERCP pancreatitis, bleeding, perforation (bile/duodenum), misplacement, migration, bile occlusion, duct abrasion, duodenal abrasion, cholangitis, severe pain) and all-death within 30 days of the index procedure.

SECONDARY ENDPOINT (Efficacy) Clinical success; normal serum bilirubin level within 14 days after onset of drainage. Relief of jaundice and pruritus.

Technical success; completion of initial ERCP and stent deployment. Procedural success; rating of stent criteria. Each criteria will be evaluated and rated as 1 for exellent, 2 for good, 3 for fair and 4 for poor.A procedure will be considered as successful if the combined rate is < 3.

Quality of life improvement by Self Assessment score at 1, 7, 14, 30, 90, 183, 274 and 365 days.

Biodegradation rate at 7, 14, 30, 90, 183, 274 and 365 days assesd by visual assessment at each follow-up visits when adequate examinations (X-ray, Endoscopy, MRI, CT, …) are performed.

Compiled Complication Rate at 7, 14, 90, 183, 274 and 365 days.

ELIGIBILITY:
Inclusion Criteria:

* 1) A subject with a biliary stricture may be entered into the study with: at least one of the following:
* Benign fibrotic distal bile duct obstruction
* Duct occlusion caused by cholelithiasis
* A benign fibrotic distal obstruction of the Common Bile Duct (CBD), demonstrated by presence of a stenosis on magnetic resonance cholangiopancreatography (MRCP) and/or ERCP with proximal ductal dilation and cholestatic liver enzymes levels
* Ductal anastomotic strictures
* Malignant Biliary stricture at least 1 cm distal to the hilum as well as periampullary hilar strictures not involving the papilla.
* Neoplasm diagnosed on clinical and imaging findings
* Post-ERCP pancreatitis
* Obstructive jaundice with evidence of pruritus, tea color urine and pale stool
* Abnormal Bilirubin rate or
* A planned exchange of plastic stents previously placed for management of symptomatic biliary stricture or
* A previous Percutaneous Transhepatic Biliary Drainage (PTBD) for management of symptomatic biliary stricture 2) Age ≥ 18 years old

Exclusion Criteria:

Patients, male or female, presenting with the following criteria may be included:

1. Subject is unwilling to comply with the follow-up schedule
2. Life expectancy < 12 m,
3. Inability to pass a guidewire through stricture
4. Contra-indication for endoscopy or interventional radiology
5. History of allergic reactions to one of the compounds of investigational product.
6. Subject is unable or refuses to give informed consent
7. Subject is pregnant or breastfeeding
8. Patient under tutorship
9. Currently participating in another trial before reaching first endpoint.
10. Pseudo Klatskin tumors (metastases in the liver hilum) and gallbladder carcinoma
11. Patient need additional biliary stenting with another device than the study device.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-16 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Safety Complication Rate for the first 30days | 30 days
  Total number of all complications is calculated as aggregate for the duration 30 days (day zero till day30 after index procedure). Two-sided 95% confidence intervals is constructed using exact (Clopper-Pearson) method.

SECONDARY OUTCOMES:
Efficacy Rates of Clinical Success | 365days
  Endpoints are analysed descriptively. Qualitative parameters are described by their distribution (frequencies and %); quantitative parameters are described by their mean, (SD±), min.-max., related to subjects with assessable data.
  Clinical Success; Normal serum bilirubin level (SBL) within 14 days after intervention. Relief of jaundice and pruritus. SBL is assessed directly before procedure day and at day14. Difference between both dates is calculated. Presence and absence of pruritus and jaundice shall behave accordingly to SBL. Postulated achieving a 20% reduction of SBL within the first 14days. Presence and absence of pruritus and jaundice is assessed and recorded at both SBL control dates.
Efficacy Rates of Technical Success | 365days
  Technical Success; Total number of completed stent deployment.

CONTACTS AND LOCATIONS:
Locations (6):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - The Prince of Wales Hospital, Hong Kong
- AIG Hospitals (Asian Institute of Gastroenterology), Hyderabad, India
- Malaysia (3):
  - Sunway Medical Centre, Kuala Lumpur
  - Universityi Kebangsaan Malaysia (UKM), Kuala Lumpur
  - University Malaya Medical Centre (UMMC)Clinical Investigation Centre (CIC), Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No